CLINICAL TRIAL: NCT01481337
Title: Prospective Observatory of Endoscopic Mucosal Colonic Resection and Polypectomy Under Aspirin : the "OPERA" Study
Brief Title: Endoscopic Mucosal Colonic Resection and Polypectomy Under Aspirin
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, VANBIERVLIET, Director, Head of Endoscopy, Principal Investigator, Medical Doctor, Société Française d'Endoscopie Digestive
Other Study IDs: OPERA
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Polyps
Keywords: colon; endoscopy; resection
MeSH Terms: conditions — Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Polypectomy or mucosal endoscopic resection under aspirin
  Interventions: Procedure: Colonic polypectomy or endoscopic mucosal resection (EMR)

INTERVENTIONS:
Procedure: Colonic polypectomy or endoscopic mucosal resection (EMR) — Resection of colonic polyps using polypectomy tehnique (with electrocoagulation) or mucosal resection (EMR or mucosectomy) with injection of physiological serum thus resection with electrocoagulation.

SUMMARY:
The endoscopic management of patients on anti platelet agents is a wide problem more and more common, with prevalence of patients on this type of therapy steadily increasing. The risk of bleeding on antiplatelet during an endoscopic examination can be major. The risk of cardiovascular thrombotic accident in dirty shutdown of anti platelet, was recently described as significant (4-5%). Current recommendations for polypectomy allow the gesture as aspirin and are based on literature data scarce, often retrospective. Such work may be for a lack of increased bleeding risk during a colonic polypectomy under aspirin. There is to date no significant data published on the implementation of the endoscopic mucosal resection (mucosectomy) under aspirin. It is necessary to achieve a national multicenter observational study on a large scale in the daily practice of colonic polypectomy / mucosectomy in patient taking aspirin.

The aim of the study is to determine the incidence of immediate and delayed bleeding colonic polypectomy and mucosectomy with aspirin. The patients undergoing colonoscopy and taking a long-term aspirin therapy and presenting a major risk of thromboembolism or medium will incluables. Inclusion will be achieved for those patients receiving aspirin colonoscopy after signing a specific consent. Polypectomy will be possible according to the recommendations of the French Society of Digestive Endoscopy. Upon discovery of a lesion to be resected by mucosectomy, the patient will benefit from the mucosectomy. The study is observational, multicenter, prospective, national. The polypectomies / colonic mucosectomies will be made using the conventional techniques and the current recommendations. The immediate and delayed hemorrhage meet specific definitional criteria. The number of patients to be included will be 1000. The duration of the study inclusions will be 36 months. The trial will be conducted in full compliance with laws, regulations and ethical aspects.

It is expected in this work that the incidence of post-polypectomy bleeding under aspirin is the same. The rate of bleeding reported in the post mucosectomy size is higher compared to the polypectomy: it is however expected that the rate of bleeding in the post mucosectomy with or without aspirin is indifferent. It will follow a recommendation of French society adapted to endoscopy for this type of procedure

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male or female
* Polypectomy AND / OR mucosectomy (EMR) performed on aspirin during a colonoscopy
* Taking a single daily dose of aspirin long-term (<375 mg for more than 3 months) in the prevention of cardiovascular and thromboembolic risk with a major or medium - secondary prevention
* Affiliation to the regime of national health protection
* Informed consent and patient's written obtained
* No participation in another clinical study

Exclusion Criteria:

* Contraindications to the achievement of a lower gastrointestinal endoscopy
* Taking a single daily dose of clopidogrel or other anti-platelet, anti vitamin K (AVK), heparin or anti bi aggregation in the context of cardiovascular prevention
* Taking chronic anti inflammatory drug (at least once weekly)
* Haemorrhagic disease, disorders of hemostasis and coagulation (PT <60%, aPTT> 40 sec. And platelets <60000/mm3), hematologic malignancy, chronic liver cirrhosis classified as Child Pugh B or C, acute or chronic renal failure
* Patient with severe disease and progressive decompensated in the opinion of the investigator
* Pregnant women, nursing
* Not signing the written consent and / or mental disabilities of the subject making its participation in the trial impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient under chronic aspirin therapy (antiplatelet agent) for cardiovascular reason who underwent colonic polypectomy or endoscopic mucosal resection.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of delayed bleeding after polypectomy and / or colonic mucosectomy (endoscopic mucosal resection) in patients on aspirin | 30 days

SECONDARY OUTCOMES:
Incidence of immediate bleeding after polypectomy and / or colonic mucosectomy in patients on aspirin | one minute
Efficacy of endoscopic hemostasis in case of bleeding induced | During the lenght of endoscopy (colonoscopy) and at 30 days
morbidity / mortality induced by immediate and delayed bleeding after polypectomy and / or colonic mucosectomy in patients on aspirin | 30 days
predictors of gastrointestinal bleeding post polypectomy / mucosectomy under aspirin by sub groups of patients obtained | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Archet 2 hospital, Nice, France